CLINICAL TRIAL: NCT06081062
Title: A Phase 3 Randomized, Double-blinded, Active-controlled, Multicenter Trial to Evaluate the Safety and Efficacy of Fabagal® (Agalsidase Beta) in Patients With Fabry Disease
Brief Title: Evaluate the Safety and Efficacy of Fabagal® (Agalsidase Beta) in Patients With Fabry Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ISU Abxis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISU303-003
Record Dates: First submitted 2023-08-08; First posted 2023-10-12 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase beta

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fabagal® (Agalsidase beta) (Experimental): 1 mg/kg, administered every 2 weeks for 12 months
  Interventions: Biological: Fabagal® (Agalsidase beta)
- Active Comparator (Agalsidase beta) (Active Comparator): 1 mg/kg, administered every 2 weeks for 12 months
  Interventions: Drug: Active comparator (Agalsidase beta)

INTERVENTIONS:
Biological: Fabagal® (Agalsidase beta) — 1 mg/kg every 2 weeks for 12 months
  Arms: Fabagal® (Agalsidase beta)
Drug: Active comparator (Agalsidase beta) — 1 mg/kg every 2 weeks for 12 months
  Arms: Active Comparator (Agalsidase beta)

SUMMARY:
Evaluate the safety and efficacy of Fabagal® developed by ISU ABXIS Co., Ltd., which has similar efficacy to active comparator (Agalsidase beta).

DETAILED DESCRIPTION:
The primary objective is to evaluate the efficacy of Fabagal compared to active comparator (Agalsidase beta). The secondary objectives will evaluate the safety, pharmacokinetics, and immunogenicity of Fabagal compared to active comparator (Agalsidase beta).

ELIGIBILITY:
Inclusion Criteria:

1. Those who have been diagnosed with Fabry disease by genetic and alpha-galactosidase A enzyme tests and grouped by sex are as follows:

   * Male: Those who have confirmed GLA mutation (variation of α-galactosidase A gene) by genetic testing, and whose activity of alpha-galactosidase A in leukocytes is 5% or less than the normal mean value
   * Female: Those who have confirmed GLA mutation by genetic testing, and whose alpha-galactosidase A is within the normal range or is deficient
2. Age: Those who are aged 8 years or older
3. Those who have at least one of the following symptoms and signs:

   * Glomerular filtration rate decreased (Inclusion criteria: 2 or more cases of 30 ≦ eGFR < 90 mL/min/1.73 m2 [adjusted for age >40] [including results within 6 months of the screening visit, but including results within 12 months for patients with a 60 ≦ eGFR < 90 mL/min/1.73 m2])

     * Proteinuria that is equivalent to microalbuminuria or worse (Inclusion criteria: 2 or more cases of creatinine 30 mg/g in random urine at least 24 hours apart [including results within 6 months of the screening visit] or ≥30 mg of albuminuria in 24-hour urine)

       * For 24 hr urinary protein extraction (>4 mg/m2/hr) or for spot urinary protein/creatinine ratio (≥200 mg/g [Cr]) *Pediatrics: Aged <19 years

         * Abnormal left ventricular function as evidenced by MRI or echocardiography

           * Left ventricular mass index (LVMI)* >115 g/m2 (male), >95 g/m2 (female) or
           * Left ventricular wall thickness >12 mm (However, in the case of patients with hypertension, patients must have blood pressure treatment for at least 6 months prior to administration of the same drug) etc.

             * Clinically significant arrhythmias and conduction disturbances, etc.

               * Stroke or transient ischemic attack, etc., as evidenced by objective testing
4. Patients who have not previously received enzyme replacement therapy (ERT) or Chaperone therapy for treatment of Fabry disease
5. Patients who voluntarily consented and signed the informed consent form
6. Patients (female patients and partners of male patients who are of childbearing potential) who have agreed to use a medically appropriate method of contraception (intrauterine device, condoms, surgical methods such as vasectomy) during the clinical study

Exclusion Criteria:

1. Patients who participated in other studies in which investigational products are administered within 30 days prior to the screening visit
2. Patients with chronic kidney disease stage 4 to 5 (CKD 4-5; see Section 16.1)
3. Patients who are currently on dialysis or have a history of kidney transplantation, or patients scheduled for dialysis at the time of screening, or waitlisted for kidney transplantation
4. Patients who have started angiotensin-converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB) treatment within 4 weeks prior to the screening visit or whose dose has been changed
5. Patients who are pregnant, breastfeeding, or planning to become pregnant or breastfeed during the clinical study
6. Patients with a history of HIV, hepatitis B/C or HIV antibodies, hepatitis B surface antigens, or hepatitis C antibodies
7. Patient whose medical, emotional, behavioral, or psychological conditions appear to interfere with compliance with the requirements of the clinical study according to the investigator's judgment

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of Fabagal compared with active comparator (Agalsidase beta) | Screening visit (Visit 0) and Visit 25 (Day 336)
  The proportion of patients achieving a GL-3 score (score 0) in renal cells after treatment with Fabagal or Active comparator (Agalsidase beta) in patients with Fabry disease
  The proportion of patients achieving a GL-3 score (score 0) in renal cells after treatment with Fabagal or Active comparator (agalsidase beta) in patients with Fabry disease The primary endpoint is a comparison of the proportion of subjects in each group who achieve a score of Zero on the renal capillary endothelium histology.
  The score is graded on a scale from 0-3 (normal, mild, moderate, and severe).
  * 0: signified no visible inclusions
  * 1: signified multiple discrete lipid granules
  * 2: signified single or multiple aggregates of lipid granules
  * 3: signified aggregates of lipid granules either large enough or numerous enough to cause clear distortion of the luminal surface

SECONDARY OUTCOMES:
Change from baseline in GL-3 levels in renal cells after administration of 24 doses of Fabagal compared to active comparator | Screening visit (Visit 0) and Visit 25 (Day 336)
  After administering Fabagal injection and active control group 24 times, changes in GL-3 levels in kidney cells compared to baseline will be confirmed.
Change from baseline in GL-3/lyso Gb-3 concentration in urine and blood after administration of 24 doses of Fabagal compared to active comparator | Screening visit (Visit 0), Visits 3, 5, 7, 9, and 11 (Days 28, 56, 84, 112, and 140), Visit 13 (Day 168), Visits 15, 17, 19, 21, and 23 (Days 196, 224, 252, 280, and 308) and Visit 25 (Day 336)
  Plasma and urine GL-3 are often elevated in the plasma of patients diagnosed with Fabry disease. After administering Fabagal injection and the active control group 24 times, the change in GL-3 and lyso Gb-3 concentrations in urine and blood compared to the baseline value will be confirmed.
Change from baseline in renal function test values (estimated Glomerular Filtration Rate, eGFR) after administration | Screening visit (Visit 0), Visit 13 (Day 168), and Visit 25 (Day 336)
  Evaluated at Screening visit (Visit 0, Baseline), Visit 13 (Day 168) and Visit 25 (Day 336). eGFR is an estimation of the glomerular filtration rate of the renal (how much blood the kidneys are filtering).
Change from baseline in pain score after administration of 24 doses of Fabagal compared to active comparator (Short Form McGill Pain Questionnaire-2) | Visits 1, 13, and 25 (Days 0, 168, and 336)
  The SF-MPQ-2 has 22 questions (6 on persistent pain, 6 on intermittent pain, 6 on neuropathic pain, and 4 on emotional pain) to be rated on an 11-point intensity scale (0 for not at all, to 10 for worst thinkable). Pain scores are presented as the mean of the ratings of all items.
Change from baseline in quality of life after administration of 24 doses of Fabagal compared to active comparator (SF-36v2 questionnaire) | Visits 1, 13, and 25 (Days 0, 168, and 336)
  The SF-36v2 consists of 36 questions(8-domain) to measure functional health and happiness from the patient's perspective. The 8 domains are physical functioning, role - physical, bodily pain, general health, vitality, social functioning, role - emotional, and mental health. The domain score is the sum of the weights of questions in each item. The score distribution ranges from 0 to 100, with a low score indicating a poor quality of life.

CONTACTS AND LOCATIONS:
Locations (3):
- Philippines (2):
  - Philippine General Hospital, Manila
  - St.Luke's Medical Center, Manila
- Seoul Asan Center, Seoul, Songpa-gu, South Korea